CLINICAL TRIAL: NCT00195650
Title: A Multi-Center Continuation Study of the Human Anti-TNF Antibody D2E7 Administered as a Subcutaneous Injection in Patients With Rheumatoid Arthritis
Brief Title: Long Term Open Label Continuation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DE020
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Open-label adalimumab 40 mg
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Subcutaneous injection of 40 mg adalimumab every other week (eow) or monthly for up to 520 weeks (10 years)
  Other Names: Humira, ABT-D2E7

SUMMARY:
The purpose of the study was to assess the long-term safety and clinical efficacy following repeated administration of adalimumab in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Study DE020 was a multicenter, open-label continuation study for patients with rheumatoid arthritis who had participated in a prior Phase 1, 2, or 3 adalimumab study in the United States or Canada, had a favorable safety and efficacy profile when treated with adalimumab, and met the eligibility criteria for the continuation study. Participants received subcutaneous injections of adalimumab every other week (eow) or monthly based on the adalimumab regimen received in the prior study (i.e., participants who received monthly dosing in the prior study began the continuation study on monthly dosing; all other participants began adalimumab dosing at eow intervals). Participants who maintained an American College of Rheumatology 50% (ACR50) response for 2 consecutive visits could have their dosing interval lengthened to a monthly dosing schedule. Safety and efficacy data were collected over 520 weeks (10 years). Both safety and efficacy data were analyzed using all participants who received at least 1 dose of open-label adalimumab in the 10-year continuation study DE020 (the Full Analysis Set, n=846). Three patients who entered the continuation study but were never dosed were excluded from all analyses.

ELIGIBILITY:
Inclusion Criteria

* Participant was in a prior D2E7 (adalimumab) study
* Participant was age 18 or older and in good health (Investigator discretion) with a recent stable medical history.

Exclusion Criteria

* Participant was considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Participant was a female subject who is pregnant or breast-feeding or considering becoming pregnant
* Participant had any ongoing chronic or active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2000-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Kupper, MD, Study Director — Abbott
Locations (92):
- United States (74):
  - Site Reference ID/Investigator# 538, Birmingham, Alabama
  - Site Reference ID/Investigator# 4111, Birmingham, Alabama
  - Site Reference ID/Investigator# 4113, Mobile, Alabama
  - Site Reference ID/Investigator# 408, Anchorage, Alaska
  - Site Reference ID/Investigator# 537, Tucson, Arizona
  - Site Reference ID/Investigator# 66822, Anaheim, California
  - Site Reference ID/Investigator# 557, La Jolla, California
  - Site Reference ID/Investigator# 387, Los Angeles, California
  - Site Reference ID/Investigator# 555, Los Angeles, California
  - Site Reference ID/Investigator# 552, Santa Barbara, California
  - Site Reference ID/Investigator# 66864, Santa Monica, California
  - Site Reference ID/Investigator# 535, Stanford, California
  - Site Reference ID/Investigator# 3412, Upland, California
  - Site Reference ID/Investigator# 451, Westlake Village, California
  - Site Reference ID/Investigator# 572, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 4109, Denver, Colorado
  - Site Reference ID/Investigator# 541, Danbury, Connecticut
  - Site Reference ID/Investigator# 654, Milford, Connecticut
  - Site Reference ID/Investigator# 655, Wilmington, Delaware
  - Site Reference ID/Investigator# 455, Daytona Beach, Florida
  - Site Reference ID/Investigator# 431, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 574, Fort Myers, Florida
  - Site Reference ID/Investigator# 66843, Gainesville, Florida
  - Site Reference ID/Investigator# 579, Orlando, Florida
  - Site Reference ID/Investigator# 571, Palm Harbor, Florida
  - Site Reference ID/Investigator# 651, Sarasota, Florida
  - Site Reference ID/Investigator# 66863, St. Petersburg, Florida
  - Site Reference ID/Investigator# 542, Tampa, Florida
  - Site Reference ID/Investigator# 415, Vero Beach, Florida
  - Site Reference ID/Investigator# 652, Zephyrhills, Florida
  - Site Reference ID/Investigator# 449, Boise, Idaho
  - Site Reference ID/Investigator# 4110, Boise, Idaho
  - Site Reference ID/Investigator# 650, Coeur d'Alene, Idaho
  - Site Reference ID/Investigator# 578, Chicago, Illinois
  - Site Reference ID/Investigator# 4112, Indianapolis, Indiana
  - Site Reference ID/Investigator# 547, Louisville, Kentucky
  - Site Reference ID/Investigator# 534, Metairie, Louisiana
  - Site Reference ID/Investigator# 544, Chevy Chase, Maryland
  - Site Reference ID/Investigator# 653, Boston, Massachusetts
  - Site Reference ID/Investigator# 4114, Worcester, Massachusetts
  - Site Reference ID/Investigator# 546, Petoskey, Michigan
  - Site Reference ID/Investigator# 577, St Louis, Missouri
  - Site Reference ID/Investigator# 549, Billings, Montana
  - Site Reference ID/Investigator# 561, Reno, Nevada
  - Site Reference ID/Investigator# 573, Dover, New Jersey
  - Site Reference ID/Investigator# 66842, Toms River, New Jersey
  - Site Reference ID/Investigator# 559, Voorhees Township, New Jersey
  - Site Reference ID/Investigator# 562, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 66823, Brooklyn, New York
  - Site Reference ID/Investigator# 432, Lake Success, New York
  - Site Reference ID/Investigator# 657, New York, New York
  - Site Reference ID/Investigator# 647, New York, New York
  - Site Reference ID/Investigator# 545, Port Jefferson Station, New York
  - Site Reference ID/Investigator# 540, Syracuse, New York
  - Site Reference ID/Investigator# 646, Statesville, North Carolina
  - Site Reference ID/Investigator# 438, Cincinnati, Ohio
  - Site Reference ID/Investigator# 436, Dayton, Ohio
  - Site Reference ID/Investigator# 548, Bend, Oregon
  - Site Reference ID/Investigator# 553, Eugene, Oregon
  - Site Reference ID/Investigator# 532, Portland, Oregon
  - Site Reference ID/Investigator# 570, Bethlehem, Pennsylvania
  - Site Reference ID/Investigator# 575, Ridley Park, Pennsylvania
  - Site Reference ID/Investigator# 585, Willow Grove, Pennsylvania
  - Site Reference ID/Investigator# 2435, Dallas, Texas
  - Site Reference ID/Investigator# 536, Richmond, Virginia
  - Site Reference ID/Investigator# 649, Everett, Washington
  - Site Reference ID/Investigator# 66862, Everett, Washington
  - Site Reference ID/Investigator# 531, Kirkland, Washington
  - Site Reference ID/Investigator# 412, Olympia, Washington
  - Site Reference ID/Investigator# 658, Spokane, Washington
  - Site Reference ID/Investigator# 576, Vancouver, Washington
  - Site Reference ID/Investigator# 551, Yakima, Washington
  - Site Reference ID/Investigator# 656, Glendale, Wisconsin
  - Site Reference ID/Investigator# 539, Milwaukee, Wisconsin
- Canada (18):
  - Site Reference ID/Investigator# 513, Calgary
  - Site Reference ID/Investigator# 568, Charlottetown
  - Site Reference ID/Investigator# 565, Hamilton
  - Site Reference ID/Investigator# 564, Hamilton
  - Site Reference ID/Investigator# 569, Kitchener
  - Site Reference ID/Investigator# 3440, Montreal
  - Site Reference ID/Investigator# 413, Montreal
  - Site Reference ID/Investigator# 66805, North York
  - Site Reference ID/Investigator# 66807, North York
  - Site Reference ID/Investigator# 414, Ottawa
  - Site Reference ID/Investigator# 566, Pointe-Claire
  - Site Reference ID/Investigator# 2467, Sainte-Foy, Quebec
  - Site Reference ID/Investigator# 66804, Scarborough
  - Site Reference ID/Investigator# 563, St. John's
  - Site Reference ID/Investigator# 2466, Toronto
  - Site Reference ID/Investigator# 567, Toronto
  - Site Reference ID/Investigator# 3442, Vancouver
  - Site Reference ID/Investigator# 514, Winnipeg

REFERENCES:
- [Derived] Furst DE, Kavanaugh A, Florentinus S, Kupper H, Karunaratne M, Birbara CA. Final 10-year effectiveness and safety results from study DE020: adalimumab treatment in patients with rheumatoid arthritis and an inadequate response to standard therapy. Rheumatology (Oxford). 2015 Dec;54(12):2188-97. doi: 10.1093/rheumatology/kev249. Epub 2015 Jul 21. PMID 26199453

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab
Started | 846 (Participants who received at least 1 adalimumab dose in study;3 enrolled did not receive adalimumab.)
Completed | 321
Not Completed | 525
Not completed — Adverse Event | 194
Not completed — Lack of Efficacy | 99
Not completed — Withdrawal by Subject | 67
Not completed — Lost to Follow-up | 44
Not completed — Death | 23
Not completed — Protocol Violation | 15
Not completed — Administrative reasons | 83

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 846
Age Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 661
  Male | 185

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting American College of Rheumatology 20% (ACR20) Response Criteria at Week 520
Description: ACR20 response criteria were: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of the 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-reactive protein (a laboratory marker of inflammation that is sensitive to acute changes in inflammatory response). All improvements were assessed relative to the baseline of the prior study.
Time Frame: Week 520
Population: All participants who received at least 1 dose of open-label adalimumab in the continuation study (Full Analysis Set) and had a Week 520 visit. Analysis used observed data (no imputation).
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 238
participants | 187

2. Primary Outcome: Number of Participants Meeting American College of Rheumatology 20% (ACR20) Response Criteria at Week 260
Description: as for outcome 1
Time Frame: Week 260
Population: All participants who received at least 1 dose of open-label adalimumab in the continuation study (Full Analysis Set) and had a Week 260 visit. Analysis used observed data (no imputation).
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 516
participants | 402

3. Primary Outcome: Number of Participants Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Week 520
Description: ACR50 response criteria were: >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of the 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-reactive protein (a laboratory marker of inflammation that is sensitive to acute changes in inflammatory response). All improvements were assessed relative to the baseline of the prior study.
Time Frame: Week 520
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 238
participants | 132

4. Secondary Outcome: Reported Adverse Events
Description: Adverse events were collected during the course of the study (after the first adalimumab injection in this continuation study DE020 through 70 days after the last adalimumab injection) for all participants who received at least 1 dose of open-label adalimumab in the continuation study (Full Analysis Set). The number of participants experiencing any adverse event (serious and non-serious) are summarized. See the Reported Adverse Events section for details.
Time Frame: Duration of study (up to 520 weeks [10 years])
Population: All participants who received at least 1 dose of open-label adalimumab in the continuation study (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 846
participants | 808

5. Primary Outcome: Number of Participants Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Week 260
Description: as for outcome 3
Time Frame: Week 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 516
participants | 279

6. Primary Outcome: Number of Participants Meeting American College of Rheumatology 70% (ACR70) Response Criteria at Week 520
Description: ACR70 response criteria were: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of the 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-reactive protein (a laboratory marker of inflammation that is sensitive to acute changes in inflammatory response). All improvements were assessed relative to the baseline of the prior study.
Time Frame: Week 520
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 238
participants | 78

7. Primary Outcome: Number of Participants Meeting American College of Rheumatology 70% (ACR70) Response Criteria at Week 260
Description: as for outcome 6
Time Frame: Week 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 516
participants | 179

8. Primary Outcome: Number of Participants in Clinical Remission (Based on Modified Disease Activity Score) at Week 520
Description: Clinical remission on modified Disease Activity Score (DAS28) was a value <2.6; >=2.6 to <=3.2 indicated low disease activity; >3.2 to <=5.1 indicated moderate disease activity; and >5.1 indicated high disease activity. DAS28 score is calculated using the number of tender joints and swollen joints (out of 28 each), patient global assessment of disease activity, and C-reactive protein (a laboratory marker of inflammation that is sensitive to acute changes in inflammatory response).
Time Frame: Week 520
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 236
participants | 135

9. Primary Outcome: Number of Participants in Clinical Remission (Based on Modified Disease Activity Score) at Week 260
Description: as for outcome 8
Time Frame: Week 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 513
participants | 243

10. Primary Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ) at Week 520
Description: The HAQ-DI is a measure of disability that ranges from 0 to 3. Decrease in score indicates improvement in physical function; a decrease of 0.22 or greater from Baseline score is clinically significant. Participants assessed their ability to perform at least 6 of the following 8 specific tasks (1. dress/groom; 2. arise; 3. eat; 4. walk; 5. reach; 6. grip; 7. maintain hygiene; 8. maintain daily activity) over the past week by marking their response on a questionnaire. Possible responses/scores included the following: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). The 8 task scores are added and the sum is divided by the number of tasks assessed (range = 6 to 8). This yields a HAQ-DI score of 0 to 3.
Time Frame: Baseline of prior Phase 1, 2, or 3 adalimumab study and Week 520
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 238
units on a scale | -0.52 (0.662)

11. Primary Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ) at Week 260
Description: as for outcome 10
Time Frame: Baseline of prior Phase 1, 2, or 3 adalimumab study and Week 260
Population: All participants who received at least 1 dose of open-label adalimumab (Full Analysis Set) in the continuation study and had a Week 260 visit. Analysis used observed data (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 515
units on a scale | -0.59 (0.628)

ADVERSE EVENTS:
Time Frame: After the first adalimumab injection in this continuation study DE020 to 70 days after the last adalimumab injection.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 432/846
Other Adverse Events (participants affected / at risk) | 768/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=846)
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Abscess limb (Infections and infestations) | 1
Abscess rupture (Infections and infestations) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myocardial infarction (Cardiac disorders) | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Adrenal insufficiency (Endocrine disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Anaemia postoperative (Injury, poisoning and procedural complications) | 2
Anaphylactic reaction (Immune system disorders) | 2
Angina pectoris (Cardiac disorders) | 14
Angina unstable (Cardiac disorders) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Antiphospholipid syndrome (Immune system disorders) | 1
Aortic aneurysm (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Appendiceal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Arrhythmia (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthritis bacterial (Infections and infestations) | 4
Arthritis infective (Infections and infestations) | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 9
Atrial flutter (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 2
Atypical mycobacterial infection (Infections and infestations) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bacteraemia (Infections and infestations) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Benign biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bradycardia (Cardiac disorders) | 3
Brain contusion (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchitis (Infections and infestations) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis viral (Infections and infestations) | 2
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Bunion (Musculoskeletal and connective tissue disorders) | 2
Bursitis infective (Infections and infestations) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 7
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Carpal tunnel syndrome (Nervous system disorders) | 1
Cellulitis (Infections and infestations) | 20
Cellulitis orbital (Infections and infestations) | 1
Cellulitis staphylococcal (Infections and infestations) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 9
Cervical cord compression (Nervous system disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Cervical myelopathy (Nervous system disorders) | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 3
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 5
Cholecystitis acute (Hepatobiliary disorders) | 4
Cholelithiasis (Hepatobiliary disorders) | 6
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Coccidioidomycosis (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colonic polyp (Gastrointestinal disorders) | 1
Colostomy closure (Surgical and medical procedures) | 1
Confusional state (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Coronary artery disease (Cardiac disorders) | 10
Coronary artery occlusion (Cardiac disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1
Cutis laxa (Skin and subcutaneous tissue disorders) | 1
Death (General disorders) | 1
Deep vein thrombosis (Vascular disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Device dislocation (General disorders) | 5
Device failure (General disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Diplopia (Eye disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 2
Diverticulitis (Infections and infestations) | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Endocarditis (Infections and infestations) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Epidural lipomatosis (Nervous system disorders) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 5
Foot operation (Surgical and medical procedures) | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 1
Gallbladder abscess (Infections and infestations) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gangrene (Infections and infestations) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastroenteritis (Infections and infestations) | 5
Gastroenteritis salmonella (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gastrointestinal infection (Infections and infestations) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Goitre (Endocrine disorders) | 4
Granuloma (General disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 1
Heart rate irregular (Investigations) | 1
Hepatic ischaemia (Hepatobiliary disorders) | 1
Herpes zoster opthalmic (Infections and infestations) | 1
Hiatus hernia, obstructive (Gastrointestinal disorders) | 2
Hip arthroplasty (Surgical and medical procedures) | 2
Hip fracture (Injury, poisoning and procedural complications) | 8
Humerus fracture (Injury, poisoning and procedural complications) | 4
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Hypertensive encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 3
Hypothyroidism (Endocrine disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7
Intestinal infarction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 2
Iron deficiency aenemia (Blood and lymphatic system disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 5
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 2
Labyrinthitis (Infections and infestations) | 1
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leg amputation (Surgical and medical procedures) | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Limb deformity (Musculoskeletal and connective tissue disorders) | 2
Lobar pneumonia (Infections and infestations) | 4
Localised infection (Infections and infestations) | 3
Loss of consciousness (Nervous system disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 7
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Lung abscess (Infections and infestations) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lyme disease (Infections and infestations) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Maculopathy (Eye disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Medical device complication (General disorders) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningitis viral (Infections and infestations) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Migraine (Nervous system disorders) | 1
Multi-organ failure (General disorders) | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 10
Myocardial ischaemia (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neck injury (Injury, poisoning and procedural complications) | 1
Necrotising fasciitis (Infections and infestations) | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephrolithiasis (Renal and urinary disorders) | 5
Nocardiosis (Infections and infestations) | 1
Nodal marginal zone B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Non-cardiac chest pain (General disorders) | 5
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Obesity (Metabolism and nutrition disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 44
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Osteomyelitis (Infections and infestations) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 2
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 5
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paresthesia (Nervous system disorders) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1
Pericardial disease (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pericarditis adhesive (Cardiac disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peritoneal tuberculosis (Infections and infestations) | 2
Peritonitis (Gastrointestinal disorders) | 1
Peritonsillar abscess (Infections and infestations) | 1
Phlebitis (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 36
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Post procedural infection (Infections and infestations) | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Postoperative wound infection (Infections and infestations) | 1
Presyncope (Nervous system disorders) | 1
Procedural complication (Injury, poisoning and procedural complications) | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1
Radiculopathy (Nervous system disorders) | 2
Rectal prolapse (Gastrointestinal disorders) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 7
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 73
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4
Sarcoidosis (Immune system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 7
Septic shock (Infections and infestations) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 5
Spinal cord compression (Nervous system disorders) | 1
Spinal decompression (Surgical and medical procedures) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Staphylococcal abscess (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 3
Staphylococcal sepsis (Infections and infestations) | 2
Stress urinary incontinence (Renal and urinary disorders) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2
Sudden death (General disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 3
Syncope (Nervous system disorders) | 5
Synovitis (Musculoskeletal and connective tissue disorders) | 3
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tachycardia (Cardiac disorders) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombosis (Vascular disorders) | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 4
Tracheobronchitis (Infections and infestations) | 1
Transient ischaemic attack (Nervous system disorders) | 7
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 5
Urosepsis (Infections and infestations) | 7
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 4
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 2
Viral infection (Infections and infestations) | 1
Vitreous haemorrhage (Eye disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
West nile viral infection (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wound infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Xerosis (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=846)
Abdominal pain (Gastrointestinal disorders) | 48
Abdominal pain upper (Gastrointestinal disorders) | 52
Alanine aminotransferase increased (Investigations) | 52
Anaemia (Blood and lymphatic system disorders) | 62
Anxiety (Psychiatric disorders) | 74
Arthralgia (Musculoskeletal and connective tissue disorders) | 118
Aspartate aminotransferase increased (Investigations) | 46
Back pain (Musculoskeletal and connective tissue disorders) | 147
Bronchitis (Infections and infestations) | 179
Bursitis (Musculoskeletal and connective tissue disorders) | 85
Cataract (Eye disorders) | 71
Constipation (Gastrointestinal disorders) | 57
Contusion (Injury, poisoning and procedural complications) | 73
Cough (Respiratory, thoracic and mediastinal disorders) | 124
Cystitis (Infections and infestations) | 46
Depression (Psychiatric disorders) | 105
Diarrhoea (Gastrointestinal disorders) | 134
Dizziness (Nervous system disorders) | 90
Dyspepsia (Gastrointestinal disorders) | 60
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54
Fall (Injury, poisoning and procedural complications) | 55
Fatigue (General disorders) | 107
Gastroenteritis viral (Infections and infestations) | 59
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 88
Headache (Nervous system disorders) | 104
Herpes zoster (Infections and infestations) | 90
Hypercholesterolaemia (Metabolism and nutrition disorders) | 76
Hyperlipidaemia (Metabolism and nutrition disorders) | 48
Hypertension (Vascular disorders) | 176
Hypoaesthesia (Nervous system disorders) | 43
Influenza (Infections and infestations) | 87
Injection site pain (General disorders) | 56
Insomnia (Psychiatric disorders) | 93
Joint injury (Injury, poisoning and procedural complications) | 49
Limb injury (Injury, poisoning and procedural complications) | 47
Localised infection (Infections and infestations) | 46
Muscle spasms (Musculoskeletal and connective tissue disorders) | 66
Muscle strain (Injury, poisoning and procedural complications) | 51
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 54
Nasopharyngitis (Infections and infestations) | 193
Nausea (Gastrointestinal disorders) | 119
Neck pain (Musculoskeletal and connective tissue disorders) | 46
Oedema peripheral (General disorders) | 91
Oral herpes (Infections and infestations) | 48
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 70
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 59
Osteoporosis (Musculoskeletal and connective tissue disorders) | 64
Pain in extremity (Musculoskeletal and connective tissue disorders) | 88
Pneumonia (Infections and infestations) | 63
Procedural pain (Injury, poisoning and procedural complications) | 65
Pyrexia (General disorders) | 46
Rash (Skin and subcutaneous tissue disorders) | 131
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 215
Sinusitis (Infections and infestations) | 211
Tooth abscess (Infections and infestations) | 49
Upper respiratory tract infection (Infections and infestations) | 392
Urinary tract infection (Infections and infestations) | 170
Vomiting (Gastrointestinal disorders) | 52
Vulvovaginal mycotic infection (Infections and infestations) | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.